CLINICAL TRIAL: NCT03293407
Title: Ventavis® (Iloprost): Evaluation of Inhaled Iloprost Effects Using the Breelib™ Nebulizer, on Clinical Outcomes and Physical Activity of Patients With Advanced Pulmonary Arterial Hypertension
Brief Title: Evaluation of Inhaled Iloprost Effects Using the Breelib Nebulizer, on Clinical Outcomes and Physical Activity of Patients With Advanced Pulmonary Arterial Hypertension
Acronym: VENTASTEP
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19398
Record Dates: First submitted 2017-09-20; First posted 2017-09-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary arterial hypertension; PAH
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Iloprost

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAYQ6256_Ventavis: Patients with pulmonary hypertension who agree to be treated with Ventavis (Iloprost) at the discretion of physician
  Interventions: Drug: Iloprost (Ventavis, BAYQ6256); Device: Breelib nebulizer

INTERVENTIONS:
Drug: Iloprost (Ventavis, BAYQ6256) — Using Breelib device
Device: Breelib nebulizer — Used for inhalation of Ventavis

SUMMARY:
The main aim of the observational VENTASTEP study was to investigate the association between changes in clinical outcome measures and changes in device outcome measures in PAH patients using the new Breelib nebulizer in a real life setting.

The study was not designed to investigate or confirm the effectiveness and safety of iloprost.

ELIGIBILITY:
Inclusion Criteria:

* Ventavis-treatment naïve patients aged ≥18 years at initiation of Ventavis (Iloprost) therapy diagnosed with pulmonary arterial hypertension WHO FC III
* Patients who are planned to be treated with Ventavis (Iloprost) and where the decision to use the Breelib has been agreed by physician and patient
* Patients who are willing to wear a smart watch (iWatch2) over the observation period of 3 months ± 2 weeks
* Signed informed consent

Exclusion Criteria:

* Patients allergic to Nickel and Methacrylates
* Patients participating in an investigational program with interventions outside of routine clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension at intermediate risk and WHO FC III who failed to respond adequately to initial therapy with one or more PAH drugs or who clinically deteriorated after initial treatment response and for whom a therapy escalation with Ventavis (Iloprost) has been agreed by patient and physician.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Change of Six-minute walking distance (6MWD) | Baseline and 3 months
  Clinical outcome measured by study nurse.
Change of laboratory results of the biomarkers NT-pro BNP/BNP | Baseline and 3 months
Change of Health related Quality of Life-EuroQol five dimensions questionnaire (EQ-5D) | Baseline and 3 months
Change of World Health Organization functional class | Baseline and 3 months
Change of Distance Walked per day | Baseline and 3 months
Change of Number of Steps per day | Baseline and 3 months
Change of number of floors climbed (10 feet) per day | Baseline and 3 months
Change of time spent at home per day | Baseline and 3 months
Change of number of relevant location changes per day | Baseline and 3 months
Change of number of times leaving home per day | Baseline and 3 months
Change of number of times standing up per day | Baseline and 3 months
Change of 6MWD | Baseline and 3 months
  Device based outcome measured by smart device.
Heart rates during baseline and observation period | Up to 3 months

SECONDARY OUTCOMES:
The average daily inhalation duration per session | Up to 3 months
The average number of daily inhalations | Up to 3 months
Change of sleep quality | Baseline and 3 months
  Measured by Pittsburgh Sleep Quality Index (PSQI).
Incidence of AEs | Up to 3 months after first inhalation
Change of heart rate during 6MWD | Baseline and 3 months
The average daily proportion of complete/incomplete inhalations | Up to 3 months
The average association between physical activity level (wearable device based) and time to last inhalation | Up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Germany

REFERENCES:
- [Background] Mueller C, Stollfuss B, Roitenberg A, Harder J, Richter MJ. Evaluation of Clinical Outcomes and Simultaneous Digital Tracking of Daily Physical Activity, Heart Rate, and Inhalation Behavior in Patients With Pulmonary Arterial Hypertension Treated With Inhaled Iloprost: Protocol for the Observational VENTASTEP Study. JMIR Res Protoc. 2019 Apr 15;8(4):e12144. doi: 10.2196/12144. PMID 30985279
- [Derived] Stollfuss B, Richter M, Dromann D, Klose H, Schwaiblmair M, Gruenig E, Ewert R, Kirchner MC, Kleinjung F, Irrgang V, Mueller C. Digital Tracking of Physical Activity, Heart Rate, and Inhalation Behavior in Patients With Pulmonary Arterial Hypertension Treated With Inhaled Iloprost: Observational Study (VENTASTEP). J Med Internet Res. 2021 Oct 8;23(10):e25163. doi: 10.2196/25163. PMID 34623313